CLINICAL TRIAL: NCT05461430
Title: Mass Response of Tumor Cells as a Biomarker for Rapid Therapy Guidance
Brief Title: Mass Response of Tumor Cells as a Biomarker for Rapid Therapy Guidance (TraveraRTGx)
Acronym: TraveraRTGx
Status: Recruiting | Type: Observational
Sponsor: Travera Inc (Industry)
Collaborators: xCures (Industry)
Responsible Party: Sponsor
Other Study IDs: TRV-003
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-11

CONDITIONS: Pleural Effusion, Malignant; Ascites, Malignant; Carcinoma; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Carcinoma, Renal; Carcinoma, Small Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Pancreatic Ductal; Carcinoma, Neuroendocrine; Carcinoma, Thymic; Carcinoma, Pancreatic; Carcinoma Breast; Carcinoma, Ovarian; Carcinoma Bladder; Carcinoma of Unknown Primary; Carcinoma of the Head and Neck; Carcinoma of the Oropharynx; Carcinoma of the Larynx; Carcinoma of the Bladder; Carcinoma of Esophagus; Carcinoma of the Nasopharynx; Carcinoma of the Penis; Carcinoma of the Cervix; Carcinoma of the Anus; Carcinoma of the Vulva; Carcinoma of the Appendix; Carcinoma of the Oral Cavity; Cholangiocarcinoma; Melanoma; Mesothelioma; Pancreatic Cancer
Keywords: Breast Cancer; Lung Cancer; NSCLC; Occult Cancer; Ovarian Cancer; Melanoma; Mesothelioma; Gastrointestinal Stromal Tumor; Gastric Cancer; Colon Cancer; Cervical Cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Ascites; Carcinoma; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Carcinoma, Small Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Pancreatic Ductal; Carcinoma, Neuroendocrine; Thymoma; Pancreatic Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Urinary Bladder Neoplasms; Neoplasms, Unknown Primary; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Esophageal Neoplasms; Nasopharyngeal Neoplasms; Penile Neoplasms; Uterine Cervical Neoplasms; Anus Neoplasms; Vulvar Neoplasms; Appendiceal Neoplasms; Mouth Neoplasms; Cholangiocarcinoma; Melanoma; Mesothelioma; Lung Neoplasms; Gastrointestinal Stromal Tumors; Stomach Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this study, sponsored by Travera Inc. in Massachusetts, is to validate whether the mass response biomarker has potential to predict response of patients to specific therapies or therapeutic combinations using isolated tumor cells from various specimen formats including malignant fluids such as pleural effusions and ascites, core needle biopsies, fine needle aspirates, or resections.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years of age
2. Written Informed Consent provided by patient
3. Diagnosis of any kind of carcinoma
4. Malignant fluid (e.g. pleural effusion or ascites) drainage OR tumor tissue resection OR tumor tissue needle biopsy is clinically indicated as part of SOC
5. Proceeding onto therapy for treatment
6. Informed consent obtained for the XCELSIOR longitudinal outcomes registry (NCT03793088)

Exclusion Criteria:

1. Lack of informed consent
2. Unable to obtain sufficient sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This pilot study will utilize samples from as many as 200 patients with a known carcinoma undergoing routine draining of malignant fluids or sampling of their tumor tissue for diagnostic or palliative standards of care (SOC).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
BOR | 12 months
  Best overall response

SECONDARY OUTCOMES:
PFS | 24 months
  Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stevens, Phd, Principal Investigator — Travera Inc; Rob Kimmerling, Phd, Principal Investigator — Travera Inc
Locations (1):
- xCures, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No